CLINICAL TRIAL: NCT02251938
Title: A Phase IIIb, Multinational, Multicenter, Open-Label Extension Study Assessing the Long-Term Safety of PRN Intravitreal Injections of DE-109 in Subjects With Non-Infectious Uveitis of the Posterior Segment of the Eye Who Have Participated in the SAKURA Development Program
Acronym: SPRING
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Santen Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 32-009
Record Dates: First submitted 2014-09-19; First posted 2014-09-29 (Estimated); Results first posted 2020-02-12 (Actual); Last update posted 2020-02-12 (Actual); Status verified 2020-01

CONDITIONS: Non-Infectious Uveitis of the Posterior Segment of the Eye
MeSH Terms: interventions — Sirolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- DE-109 Sirolimus (Experimental): DE-109 440 μg
  Interventions: Drug: DE-109 440 μg

INTERVENTIONS:
Drug: DE-109 440 μg — Medium Dose
  Other Names: Sirolimus

SUMMARY:
The objective of this extension study is to evaluate the long-term safety of treatment with DE-109 (440 μg) in subjects with non-infectious uveitis of the posterior segment of the eye who have participated in the SAKURA development program.

DETAILED DESCRIPTION:
This is a multicenter, open-label, extension study of intravitreal injections of the 440 μg dose of DE-109 in subjects with non-infectious uveitis of the posterior segment who received any dose of DE-109 and exited the SAKURA program under Santen Protocol 32-007, Amendment 05.

Subjects who were randomized and received at least two injections of DE-109 during the first five months of the SAKURA program and obtained clinical benefit from the study medication, as determined by the Investigator, may be considered for entry in this 12-month extension study. The minimum time lag from last injection in the SAKURA program to entry into the current protocol is 60 days.

ELIGIBILITY:
Inclusion Criteria:

1. Participated in the SAKURA study
2. Received clinical benefit from treatment in the SAKURA study
3. Ability to sign informed consent and attend all study visits

Exclusion Criteria:

1. Uveitis of infectious etiology
2. Implanted device
3. Suspected or confirmed central nervous system or ocular lymphoma
4. Uncontrolled glaucoma
5. Significant ocular disease
6. Intravitreal injections in the past 60 days
7. Intraocular surgery or treatment
8. Ocular or periocular infection
9. History of herpetic infection
10. Toxoplasmosis or toxoplasmosis scar
11. Ocular malignancy
12. Vitrectomy
13. Allergy or hypersensitivity to study drug
14. Participation in other uveitis device clinical trials within 30 days
15. Any recent systemic condition/infection
16. Immunosuppressive therapy or immunocomprimised
17. Cytomegalovirus infection
18. Malignancy in remission
19. Females who are pregnant or lactating and who are not using adequate contraceptive
20. Medical marijuana or illegal drug use
21. Systemic saroidosis
22. Therapeutic radiation to the head or neck

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2014-09-29 (Actual); Primary Completion 2017-11-01 (Actual); Study Completion 2017-11-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lanita Scott, MD, Study Director — Santen Inc.
Locations (25):
- United States (13):
  - Phoenix, Arizona
  - Sacramento, California
  - Golden, Colorado
  - Tampa, Florida
  - Oak Park, Illinois
  - Jackson, Michigan
  - St Louis, Missouri
  - New Brunswick, New Jersey
  - Palisades Park, New Jersey
  - New York, New York
  - Orchard Park, New York
  - Austin, Texas
  - Salt Lake City, Utah
- Graz, Austria
- Paris, France
- India (7):
  - Hyderabad, Andhra Pradesh
  - Aurobindo Marg, New Dehli
  - Daryāganj, New Dehli
  - Bhubaneswar, Odisha
  - Chennai, Tamil Nadu
  - Madurai, Tamil Nadu
  - Noida, Uttar Pradesh
- Milan, Italy
- Turkey (Türkiye) (2):
  - Ankara
  - Izmir

RESULTS

PARTICIPANT FLOW:
Groups:
- DE-109 440 μg: Medium dose of DE-109
Period: Overall Study
Arm/Group | DE-109 440 μg
Started | 60
Completed | 43
Not Completed | 17

BASELINE CHARACTERISTICS:
Arm/Group | DE-109 440 μg
Number analyzed (Participants) | 60
Age, Continuous [Mean (Standard Deviation); unit: years] | 43.31 (15.092)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 31
  Male | 29
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 21
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 4
  White | 30
  More than one race | 2
  Unknown or Not Reported | 2
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic or Latino | 10
  Not Hispanic or Latino | 47
  Not reported | 3
Geographic Region [Count of Participants; unit: Participants]
  United States | 33
  India | 17
  Europe, the Middle East and Africa | 10

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Best Corrected Visual Acuity (BCVA) at Month 12 in the Study Eye
Description: Best Corrected Visual Acuity (BCVA) measures the acuteness or clearness of best-corrected vision in ETDRS (Early Treatment of Diabetic Retinopathy Study) letters. An increase in BCVA indicates improvement in the best-corrected vision. A BCVA score of 85 ETDRS letters is equivalent to 20/20 vision, which is considered normal vision.
Time Frame: Day 1 (Baseline) and Month 12 or early termination visit
Measure: Mean (Standard Deviation); unit: ETDRS Letters
Arm/Group | DE-109 440 μg
Number analyzed (Participants) | 43
ETDRS Letters | 2.1 (11.35)

2. Primary Outcome: Mean Change From Baseline in Intraocular Pressure at Month 12 in the Study Eye
Description: Intraocular pressure (IOP), the fluid pressure inside the eye, was measured by applanation tonometry in millimeters mercury (mmHg) with one decimal point.
Time Frame: Day 1 (Baseline) and Month 12 or early termination visit
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | DE-109 440 μg
Number analyzed (Participants) | 43
mmHg | 0.3 (4.16)

3. Primary Outcome: Number of Subjects With a Shift in Choroid Status at Month 12 in the Study Eye.
Description: Ophthalmoscopy findings were reported as normal or abnormal.
Time Frame: Day 1 (Baseline) and Month 12 or early termination visit
Measure: Number; unit: Subjects
Arm/Group | DE-109 440 μg
Number analyzed (Participants) | 43
Subjects
  Normal to Normal | 36
  Normal to Abnormal | 0
  Abnormal to Normal | 4
  Abnormal to Abnormal | 3

4. Primary Outcome: Changes From Baseline in Vitreous Haze (VH) Scores at Month 12
Description: Vitreous Haze (VH) scores were measured using the modified Standardized Uveitis Nomenclature Photographic Scale (SUN) :
  0 No inflammation
  0.5+ Trace Inflammation (slight blurring of the optic disc margins and or loss of nerve fiber layer reflex)
  1. Mild blurring of the retinal vessels and optic nerve
     1.5+ Optic nerve head and posterior retina view obstruction greater than 1+ but less than 2+
  2. Moderate blurring of the optic nerve head
  3. Marked blurring of the optic nerve head
  4. Optic Nerve head not visible
Time Frame: Day 1 (Baseline) and Month 12 or early termination visit
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | DE-109 440 μg
Number analyzed (Participants) | 43
score on a scale | -0.09 (0.847)

5. Primary Outcome: Number of Subjects Who Receive Rescue Therapy.
Description: Rescue therapy was defined as any treatment that would have a therapeutic effect on the uveitis in the posterior segment (e.g., systemic treatment with an immunosuppressant agent, or a corticosteroid injection in the study eye) other than intravitreal DE-109 determined by the Investigator.
Time Frame: By Month12
Measure: Count of Participants; unit: Participants
Arm/Group | DE-109 440 μg
Number analyzed (Participants) | 60
Participants | 9

6. Primary Outcome: Number of Subjects With a Shift in Macula Status at Month 12 in the Study Eye.
Description: Ophthalmoscopy findings were reported as normal or abnormal.
Time Frame: Day 1 (Baseline) and Month 12 or early termination visit
Measure: Number; unit: Subjects
Arm/Group | DE-109 440 μg
Number analyzed (Participants) | 43
Subjects
  Normal to Normal | 20
  Normal to Abnormal | 2
  Abnormal to Normal | 6
  Abnormal to Abnormal | 15

7. Primary Outcome: Number of Subjects With a Shift in Optic Nerve Status at Month 12 in the Study Eye.
Description: Ophthalmoscopy findings were reported as normal or abnormal.
Time Frame: Day 1 (Baseline) and Month 12 or early termination visit
Measure: Number; unit: Subjects
Arm/Group | DE-109 440 μg
Number analyzed (Participants) | 43
Subjects
  Normal to Normal | 39
  Normal to Abnormal | 2
  Abnormal to Normal | 0
  Abnormal to Abnormal | 2

8. Primary Outcome: Number of Subjects With a Shift in Retina Status at Month 12 in the Study Eye.
Description: Ophthalmoscopy findings were reported as normal or abnormal.
Time Frame: Day 1 (Baseline) and Month 12 or early termination visit
Measure: Number; unit: Subjects
Arm/Group | DE-109 440 μg
Number analyzed (Participants) | 43
Subjects
  Normal to Normal | 34
  Normal to Abnormal | 2
  Abnormal to Normal | 1
  Abnormal to Abnormal | 6

ADVERSE EVENTS:
Time Frame: An on-study Adverse Events (AEs) were collected after the date of the written informed consent until the Last Study Visit at Month 12 or early termination visit.
Groups:
- DE-109 440 μg: Medium dose of DE-109
  DE-109: Medium Dose of DE-109
Arm/Group | DE-109 440 μg
All-Cause Mortality (participants affected / at risk) | 0/60
Serious Adverse Events (participants affected / at risk) | 8/60
Other Adverse Events (participants affected / at risk) | 35/60
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | DE-109 440 μg (N=60)
Cataract (Eye disorders) | 1 (1)
Visual Acuity Reduced (Eye disorders) | 1 (1)
Vitreous Hemorrhage (Eye disorders) | 1 (1)
Intraocular Pressure Increased (Investigations) | 2 (2)
Cerebrovascular Accident (Nervous system disorders) | 1 (1)
Trigeminal Neuralgia (Nervous system disorders) | 1 (1)
Cellulitis Gangrenous (Infections and infestations) | 1 (1)
Procedural Complication (Injury, poisoning and procedural complications) | 1 (1)
Pathological Fracture (Musculoskeletal and connective tissue disorders) | 1 (1)
Lung Adenocarcinoma Metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Arterial Occlusive Disease (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | DE-109 440 μg (N=60)
Uveitis (Eye disorders) | 8 (16)
Cystoid Macular Oedema (Eye disorders) | 6 (9)
Intermediate Uvei (Eye disorders) | 6 (12)
Iridocyclitis (Eye disorders) | 3 (3)
Macular Fibrosis (Eye disorders) | 3 (4)
Intraocular Pressure Increased (Investigations) | 7 (9)
Intraocular Pressure Decreased (Investigations) | 3 (5)
Sinusitis (Infections and infestations) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2014-06-30): https://cdn.clinicaltrials.gov/large-docs/38/NCT02251938/Prot_000.pdf
  • Statistical Analysis Plan (2017-11-15): https://cdn.clinicaltrials.gov/large-docs/38/NCT02251938/SAP_001.pdf